CLINICAL TRIAL: NCT02768532
Title: VEDO-PREDIRESP Project: Value of Pharmacokinetic Assays (Vedolizumab and Anti-vedolizumab Antibody) in the Prediction of Induction and Maintenance Therapeutic Response in Crohn's Disease
Brief Title: Value of Pharmacokinetic Assays in the Prediction of Induction and Maintenance Therapeutic Response in Crohn's Disease
Acronym: VEDO-PREDIRESP
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: low inclusion rates
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Theradiag (Other); Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1608051; 2016-001587-11 (EudraCT Number)
Record Dates: First submitted 2016-05-02; First posted 2016-05-11 (Estimated); Last update posted 2023-06-15 (Actual); Status verified 2023-02

CONDITIONS: Crohn Disease
Keywords: Crohn's disease; Vedolizumab; TNF (Tumor Necrosis Factor); Clinical response; Clinical remission
MeSH Terms: conditions — Crohn Disease | interventions — vedolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Crohn's disease patients (Experimental): The patients will receive vedolizumab in compliance with the marketing authorization regimen (300 mg at weeks 0, 2, 6 and then every 8 weeks) in Crohn's Disease patients in clinical failure or intolerant to anti-TNF (Tumor Necrosis Factor) drugs. In case of lack of clinical response at week 10 or loss of response in the follow-up, all patients will be optimized with vedolizumab 300 mg at week 10 (additional infusion) and every following 4 weeks in contrast with responder patients at week 10 who will not have vedolizumab infusion at this time-point but will receive the next vedolizumab infusion at week 14 and then every 8 weeks, as recommended.
  Interventions: Drug: Vedolizumab

INTERVENTIONS:
Drug: Vedolizumab — During each 8 visits (screening, V0, V1, V2, V3, V4, V5, V6) at weeks-1, 0, 2, 6, 10, 14, 22, 54, respectively), the following parameters will be systematically recorded: Crohn's disease Activity Index (CDAI), adverse events.
  Blood and fecal samples will be systematically collected at weeks 0, 2, 6, 10, 14, 22 and 54 for routine serum ultrasensitive CRP (C-Reactive Protein) and fecal calprotectin assessments and for vedolizumab pharmacokinetic parameters, including the vedolizumab trough levels and the specific anti-Vedolizumab antibodies. In case of loss of response, an additional measurement of serum CRP (C-Reactive Protein), fecal calprotectin and Vedolizumab pharmacologic parameters will be performed.
  Other Names: Entyvio

SUMMARY:
Vedolizumab (VDZ) is a monoclonal antibody which has shown its efficacy in Crohn's disease by inducing and maintaining clinical response/remission. The French marketing authorization was obtained for Crohn's disease in patients in failure with anti-TNF (Tumor Necrosis Factor) agents.

For Crohn's disease patients treated with vedolizumab, a strong association between vedolizumab serum levels and clinical response to induction and maintenance was demonstrated by anterior studies.

It could be of paramount interest to early identify Crohn's Disease patients under vedolizumab who will be responders to vedolizumab induction and to identify those who will achieve clinical remission under maintenance therapy with vedolizumab.

Researchers decided to assess the clinical response to vedolizumab induction at week 10. For clinically non-responders at week 10, an additional dose of 300 mg of vedolizumab will be infused at week 10 and then every four weeks.

DETAILED DESCRIPTION:
Vedolizumab (VDZ) is a monoclonal antibody that binds to the heterodimer alpha 4 beta 7 integrin and which has shown its efficacy in Crohn's disease by inducing and maintaining clinical response/remission. The French marketing authorization was obtained for Crohn's disease in patients in failure with anti-TNF (Tumor Necrosis Factor) agents.

For Crohn's disease patients treated with vedolizumab, a strong association between vedolizumab serum levels and clinical response to induction and maintenance was demonstrated by anterior studies.

It could be of paramount interest to early identify Crohn's Disease patients under vedolizumab who will be responders to vedolizumab induction and to identify those who will achieve clinical remission under maintenance therapy with vedolizumab.

Researchers decided to assess the clinical response to vedolizumab induction at week 10, as the Gemini III trial has reported, among patients who had experienced previous TNF (Tumor Necrosis Factor) antagonist failure. 15% of those given vedolizumab were in remission at week 6 (P=0.433) versus 12% under placebo. At week 10, 26% under vedolizumab were in remission versus 12% in the placebo arm.

Moreover, at week 10, the proportion of patients presenting a clinical response was significantly higher in Crohn's Disease patients treated with vedolizumab (46% vs 24%).

In this study, for clinically non-responders at week 10, an additional dose of 300 mg of vedolizumab will be infused at week 10 and then every four weeks. In a post hoc analysis of GEMINI 2, additional dose of vedolizumab in patients clinically non responders to vedolizumab obtained a clinical remission in 33% of case.

ELIGIBILITY:
Inclusion Criteria :

* Aged over 18 years
* Men or non-pregnant women
* Patients with a diagnosis of Crohn's disease who requires to start Vedolizumab
* Crohn's disease defined as a Crohn's disease Activity Index (CDAI) > 150 points and/or fecal calprotectin levels > 250 µg/g of stool
* Crohn's Disease patients with previous failure with TNF (Tumor Necrosis Factor) antagonist agents and unacceptable side-effects from steroids, and/or immunosuppressive agents (i.e., azathioprine, 6-mercaptopurine, or methotrexate). In France, Vedolizumab has to be prescribed only in patients in failure or intolerant to anti-TNF.
* Patient taking corticosteroids orally, concomitant immunosuppressive agents, mesalamine, and antibiotics are allowed at stable dose for at least three months before inclusion. Steroid tapering has to be set up at Week 10 after starting Vedolizumab, according to the European Crohn and Colitis Organisation (ECCO) recommendations with a progressive decrease of steroids of 5 mg/day every week until complete withdrawn.
* Informed written consent given.

Exclusion Criteria:

* Existing pregnancy, lactation, or intended pregnancy within the next 15 months
* Minors or History of disease, including mental/emotional disorder that might interfere with their participation in the study
* Serious secondary illnesses of an acute or chronic nature, which in the opinion of the investigator renders the patient unsuitable for inclusion into the study
* Inability to comply with the protocol requirements
* Inability to fill in the diary cards during the last 7 days before each visit
* Presence of an ileo-/colonic stoma
* Patients with known colonic stricture and exclusive or predominant anal or perineal Crohn's disease lesions
* Known previous or concurrent malignancy (other than that considered surgically cured, with no evidence for recurrence for 5 years)
* Short bowel syndrome
* Previous treatments with natalizumab, efalizumab or rituximab.
* Prior extensive colonic resection, obstructive (symptomatic) intestinal stricture, abdominal abscess, active or latent tuberculosis,
* Documented Clostridium difficile superinfection;
* Indeterminate colitis
* Concomitant leukocyte apheresis.
* Any contraindication to vedolizumab therapy
* Patients who denied the protocol, not ability to accept or sign consent of the protocol
* Subject involved in another interventional clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2022-01-11 (Actual); Study Completion 2023-01-23 (Actual)

PRIMARY OUTCOMES:
Vedolizumab concentration at week 6 | Week 6
  The primary objective is to determine the optimal threshold of Vedolizumab serum concentration measured at week 6 capable to predict the clinical response at week 10 with Vedolizumab.

SECONDARY OUTCOMES:
Vedolizumab concentration at week 14 | Week 14
  Determine the optimal threshold of Vedolizumab serum concentration measured at week 14 capable to predict the clinical remission at week 54 with Vedolizumab.
Concentration of Vedolizumab at week 2 | Week 2
  Investigating whether the Vedolizumab concentrations measured at week 2 are predictive of a clinical response and clinical remission at week 10.
Presence of specific antibodies (anti-integrins) at week 2 | Week 2
  Investigating whether the presence of specific antibodies (anti-integrins) measured at week 2 are predictive of a clinical response and clinical remission at week 10.
Concentration of Vedolizumab at week 14 | Week 14
  Investigating whether the Vedolizumab concentrations measured at week 14 are predictive of a clinical response and clinical remission at week 54.
Presence of specific antibodies (anti-integrins) at week 14 | Week 14
  Investigating whether the presence of specific antibodies (anti-integrins) measured at week 14 are predictive of a clinical response and clinical remission at week 54.
Vedolizumab and calprotectin levels at week 2 | Week 2
  Analyzing the value of Vedolizumab trough levels measured at week 2 to predict a subsequent normalization of fecal calprotectin levels (< 250 micro grams/gram of stools) at week 10 under induction therapy with Vedolizumab in Crohn's Disease.
Vedolizumab and calprotectin levels at week 14 | Week 14
  Analyzing the value of Vedolizumab trough levels measured at week 14 to predict a subsequent normalization of fecal calprotectin levels (< 250 micro grams/gram of stools) at week 54 under maintenance therapy with Vedolizumab in Crohn's Disease.
Intra and inter-individual heterogeneity of Vedolizumab levels | Week 54
  Investigating the intra and inter-individual heterogeneity of Vedolizumab levels within the time-course of Vedolizumab therapy, including the induction and maintenance phases. The dosage of Vedolizumab in patients blood will be used.
Proportion of loss of clinical response | Week 54
  Comparing the proportion of loss of clinical response in responder Crohn's Disease patients as well as in primary non-responders requiring Vedolizumab dose-intensification within one-year of follow-up.
Vedolizumab serum levels | Week 54
  Comparing the Vedolizumab serum levels prior and after Vedolizumab optimization in primary non-responder patients or experiencing a loss of response (secondary non-response) requiring additional infusions of Vedolizumab.
Concentration of Vedolizumab at week 54 | Week 54
  Comparing the level of Vedolizumab between patients achieving a clinical remission or not at week 54.
Specific antibodies (anti-integrins) level at week 54 | Week 54
  Comparing the specific antibodies (anti-integrins) levels between patients achieving a clinical remission or not at week 54.

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Roblin, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (5):
- France (5):
  - CHU Kremlin Bicetre, Paris, Le Kremlin-Bicêtre
  - CHU d'Amiens, Amiens
  - CHU L'Archet, Nice
  - CHU Lyon-Sud, Hospices Civils de Lyon, PIERRE-BENITE, Pierre-Bénite
  - Chu Saint Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No